CLINICAL TRIAL: NCT01437345
Title: A Multicenter Collaborative Study on the Clinical Features, Expression Profiling, and Quality of Life of Infantile Onset Facioscapulohumeral Muscular Dystrophy
Brief Title: A Multicenter Collaborative Study on the Clinical Features, Expression Profiling, and Quality of Life of Infantile Onset FSHD
Acronym: FSHD
Status: Completed | Type: Observational
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: FSH Society, Inc. (Industry); FSHD Global Research Foundation (Other); Muscular Dystrophy Canada (Other); aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ACH0311
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for DNA and RNA analysis are optional.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is an observational study that aims to advance our knowledge on infantile onset FSHD. The study will include 50 participants of all ages who have presented with symptoms of FSHD between birth and 10 years of age. Study participation will involve a single day of assessments at one of the participating CINRG centers (to include physical exam, cognitive testing, eye exam, hearing test, strength testing and speech evaluations). The procedures may be split over additional days for scheduling purposes.

ELIGIBILITY:
Inclusion Criteria:

Affected participants must have a clinical diagnosis of FSHD, including the presence of all of the following features based on review of medical records and/or direct examination:

* Onset of symptoms involving the facial or shoulder girdle muscles
* Autosomal dominant inheritance in familial cases
* Contraction of the D4Z4 repeat array from 1-10 (10 - 38 kb) copies in the 4q35 subtelomeric region, based on established molecular genetic techniques

Exclusion Criteria:

* Symptomatic cardiomyopathy or severe cardiac arrhythmia which may limit the ability to complete the study protocol
* Maternal/mitochondrial mode of inheritance
* Evidence of an alternative diagnosis based on muscle biopsy or other available investigations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with infantile onset (diagnosed at birth until 10 years of age) and genetically confirmed FSHD will be recruited. This will include children and youth (less than 18 years old) with FSHD who are currently followed in pediatric neuromuscular centers, as well as adults (18 years or older) with FSHD who are identified as having infantile onset of disease by chart review, clinical exam, and genetic confirmation.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-07; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
All Outcome Measures | Dec 2014
  1. Establish a standardized muscle testing protocol including both manual and quantitative muscle testing as well as function testing for use in children and adults with infantile onset FSHD.
  2. To describe the clinical phenotypes of infantile FSHD; separately in the early infantile group (onset before age 5) and late onset group (onset between 5 and 10 years of age).
  3. To evaluate the impact of physical impairment, secondary health conditions, activity limitations and disability caused by FSHD on health-related quality of life and disability across different age groups; as well as to evaluate the utility of the FSHD clinical severity scale.
  4. To evaluate potential genetic modifiers of clinical phenotypes and disease progression in infantile FSHD.

CONTACTS AND LOCATIONS:
Overall Officials: Jean K Mah, MD, MS, Principal Investigator — Alberta Children's Hospital
Locations (12):
- United States (7):
  - University of California - Davis, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Children's Hospital, Durham, North Carolina
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
- Australia (2):
  - Royal Children's Hospital, Melborne
  - The Children's Hospital at Westmead, Sydney
- Alberta Children's Hospital, Calgary, Alberta, Canada
- Queen Silvia Children's Hospital, Gothenburg, Sweden
- Newcastle University, Newcastle upon Tyne, United Kingdom